CLINICAL TRIAL: NCT03913312
Title: Multicenter, One-arm, Phase II Clinical Study of Decitabine Combined With Unrelated Cord Blood Transplantation for the Treatment of Acute Myeloid Leukemia (AML) in the Elderly
Brief Title: Decitabine Combined With Unrelated Cord Blood Transplantation for Elderly Patients With AML
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Navy General Hospital, Beijing (Other); Beijing Jishuitan Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Luoyang Central Hospital (Other); People's Hospital of Zhengzhou University (Other); Dongguan People's Hospital (Other Government); The First Affiliated Hospital of Xiamen University (Other); Taian City Central Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other)
Responsible Party: Principal Investigator, Li Junmin, Director of the hematology department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-AML 2018
Record Dates: First submitted 2019-04-11; First posted 2019-04-12 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML,Elderly patients,Decitabine,Unrelated cord blood
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DAC combined with unrelated cord blood transplantation (Experimental): Decitabine (DAC) 15mg/m2/d, d-7 to d-3;Ara-C 1000g/m2/q12h, d-2 to d-1.Single unrelated cord blood (TNC>1.5*107/kg), d0.
  Interventions: Biological: Unrelated cord blood

INTERVENTIONS:
Biological: Unrelated cord blood — Unrelated cord blood comes from Shandong cord blood bank. TNC>1.5*107/kg;HLA 4-5/6

SUMMARY:
Acute myeloid leukemia (AML) is a clonal disease caused by genetic mutations in Hematopoietic stem progenitor cells. Unfortunately, advanced age (>60 years old) is considered to be one of the most important adverse prognostic factors for AML, and older patients are unable to tolerate high-dose chemotherapy, due to various complications and organ dysfunction. Based on the results of the previous research, we will carry out the pretreatment regimen of decitabine + cytarabine in elderly patients with AML who have achieved disease treatment through induction therapy, and continue the transplantation program of unrelated-blood cord blood. By assessing the patient's DFS,OS,RFS and safety to determine whether the regimen is suitable for the consolidation treatment of elderly acute myeloid leukemia, further clarify the efficacy of this regimen compared with traditional consolidation therapy, and initially confirm the effect of combined with unrelated cord blood transplantation in the treatment of acute myeloid leukemia.

DETAILED DESCRIPTION:
A prospective,Multicenter,open,single-arm clinical study.The research process is divided into three phases: the screening phase, the treatment phase, and the follow-up phase. The treatment phase includes pre-transplant pretreatment, cord blood transplantation, and consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. AML patients diagnosed by bone marrow morphology and Immunology;
2. Exclusion of APL by Bone marrow morphology or molecular level;
3. A patient who has obtained bone marrow cytology remission after inductive treatment;
4. Aged from 60 to 75 years;
5. Liver and kidney function: blood bilirubin ≤ 35μmol / L, AST or/ALT <2 times the upper limit of normal (ULN), serum creatinine;≤ 150μmol / L;
6. The function of Heart is normal;
7. Physical condition score 0-2 (ECOG score);
8. Get informed consent signed by patient or family member.

Exclusion Criteria:

1. APL patients, treatment-related AML;
2. Retreatment of patients;
3. Allergies to any of the drugs involved in the protocol;
4. There are obvious contraindications to chemotherapy drugs;
5. Liver and kidney function is obviously abnormal, exceeding the inclusion criteria;
6. Serious heart disease, including myocardial infarction, cardiac insufficiency;
7. Suffering from other organ malignant tumors at the same time ;
8. Active period of tuberculosis patients and HIV-positive patients;
9. Suffering from other blood system diseases at the same time;
10. Pregnancy or breastfeeding;
11. Cannot understand or follow the research plan;
12. A history of intolerance or allergies to similar drugs;
13. Patients under 60 years of age or over 75 years of age;
14. Participate in other clinical researchers at the same time;
15. There are other situations that hinder the conduct of the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Three years

SECONDARY OUTCOMES:
Overall Survival (OS) | Three years
  The time from enrollment to death for any reason
Complete Remission Rate (CR) | Three years
  The proportion of cases of hematologic remission that reached the total
Adverse Events (refer to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03). | Three years
  Safety/Toxicity Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Junmin Li, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiaotong University
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China